CLINICAL TRIAL: NCT03906370
Title: The Association Between Capillary Dysfunction and CD46 Phenotype in Early Diagnosed MS Patients
Brief Title: Capillary Dysfunction and CD46-immunoreceptor (CD46) Type in MS
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: MS_CD46_MRI
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples and Spinal fluid samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MS patients/cases: Patients admitted for diagnostic investigations to the MS clinic were offered participation if aged >18 years and no previous use of immunosuppressing or modifying drugs within 6 months. The diagnosis healthy/diseased was made by 2017 Mc Donald criteria.
  Interventions: Diagnostic Test: Diagnostic criteria for MS
- Healthy subjects/controls: Patients admitted for diagnostic investigations to the MS clinic were offered participation if aged >18 years and no previous use of immunosuppressing or modifying drugs within 6 months. The diagnosis healthy/diseased was made by 2017 Mc Donald criteria.

INTERVENTIONS:
Diagnostic Test: Diagnostic criteria for MS — The diagnosis healthy/diseased was made by 2017 Mc Donald criteria.
  Groups: MS patients/cases

SUMMARY:
This project aims to contribute knowledge to early MS disease mechanisms at the brain-blood interface using a combined immunological and neuroimaging approach.

The aim is to provide a novel vascular model to assess MS disease activity, and to explore its potential as an early diagnostic biomarker, prior to blood-brain barrier disruption. Additionally, the investigators want to investigate influence of immune receptor defects upon disease activity and MS brain vascular system. These aims are addressed by investigating immune receptor signals and vascular imaging modalities acquired in newly diagnosed untreated MS cohort, followed at our institution.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is considered a virus-mediated autoimmune disease in the central nerve system characterized by blood brain barrier (BBB) disruption. Conventional magnetic resonance imaging (MRI) is currently an invaluable diagnostic tool as structural lesions are accepted biomarkers. However, MRI lesions correlate poorly with disease burden underlining the clinical-radiological paradox. Therefore, more advanced MRI are needed to provide additional information beyond what is obtainable from conventional scans. Perfusion MRI alterations preceding overt BBB disruption and lesions have been described suggesting a microvascular pathology as an etiological contributor to MS lesions. Transient diffusion decrease observed by diffusion MRI support the hypothesis of a hypoxic event prior to BBB disruption. A new model of perfusion MRI (DSC) enables microvascular function assessment in MS. This model is yet to be tested on MS patients. Furthermore, emerging evidence suggest that virus receptor CD46 affects immunologic susceptibility to MS. CD46 is highly expressed on cerebral vascular endothelium and may protect BBB integrity.

The hypothesis for this project is that CD46 activity is modulator of MS disease development, where CD46 modifications increases vulnerability to BBB disruption by attenuation of normal flow responses in MS brains.

Aims: Besides testing correlations between microvascular dysfunction and MS clinical outcome, this have prompted the investigators to investigate DSC-metric and predicted microvascular dysfunction in relation to defective CD46-driven immune responses.

Method: For this the investigators conducted our MRI study performed in a clinical research setting, and the - immunological study performed in a laboratory setting. Both studies are based on newly diagnosed MS patient assessments conducted at Department of Neurology, Aarhus University Hospital. All subjects undergo clinical examination, blood/cerebrospinal fluid samples and a comprehensive 3Tesla (3T) MRI protocol. MRI parameters and immune responses are compared between study groups and related to clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 years Patients suspected with MS.

Exclusion Criteria:

Pregnancy. Drug/alcohol abuse. Cerebral tumor. Previous head injury. Previous use of immunosuppressing or modifying treatment within 6 months. Contraindications against contrast media. Baseline image analysis not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited consecutively on admission for diagnostic investigations to the MS clinic, Department of Neurology, Aarhus University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Capillary dysfunction | Baseline
  DSC- metric
CD46 dysfunction | Baseline
  CD46 immune receptor phenotype and function

CONTACTS AND LOCATIONS:
Overall Officials: Linda Sundvall, MD, Principal Investigator — Department of Neurology, Aarhus University Hospital
Locations (1):
- Department of Neurology, Aarhus, Denmark